CLINICAL TRIAL: NCT05166005
Title: The Effect of Vitamin D Supplementation in Standard Therapy on Reducing Severity of COVID-19 Among Hospitalized Patients
Brief Title: Severity of COVID-19 and Vitamin D Supplementation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitaD-COVID
Record Dates: First submitted 2021-12-12; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Respiratory Infection
Keywords: level of 25-hydroxyvitamin; 25(OH)D; vitamin D; COVID-19; treatment; prevention
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose (Active Comparator): High dose Vitamin D therapy will initiate at a dosage of 50,000 IU on the first and second week of hospitalization
  Interventions: Drug: vitamin D
- Low dose (Placebo Comparator): Vitamin D therapy will prescribe at a dosage of 2,000 IU/day
  Interventions: Drug: vitamin D

INTERVENTIONS:
Drug: vitamin D — Patients will be randomised to receive either high dose vitamin D (50,000 IU weekly) on the first and second week or low dose vitamin D (2,000 IU daily).

SUMMARY:
Purpose of the study: to analyze the interlinks between serum 25(OH)D level and severity of new coronavirus infection (COVID-19) in hospitalized patients, as well as the effect of adding colecaciferol to standard therapy for patients in the acute period of the disease.

The study will involve at least 300 hospitalized patients with confirmed COVID-19. All study participants will be twice assessed for serum 25 (OH) D levels: baseline and 8-10 days of hospitalization. Following a baseline examination, patients will be randomized into 2 groups. Group I (No. 1), vitamin D therapy begins with a dosage of 50,000 IU in the first and second weeks. Group II (No. 2), vitamin D therapy is prescribed at a dosage of 2000 IU / day. On 8-10 days of vitamin D supplementation, all participants will be retested for serum 25 (OH) D levels to assess the effectiveness of therapy. On 14-21 days we assessed severity of the course, ICU hospitalization, duration of hospitalization, outcome of the disease, duration of glucocorticoid therapy, the need for specific therapy (inhibitors IL-6), changes in cytokine/chemokine, APPs concentration.

DETAILED DESCRIPTION:
The COVID-19 pandemic that swept the world in 2019 radically changed not only the social sphere of life, subordinating everything around to its influence, but also the healthcare sector. It affected both its practical and scientific sides, globally changing the approach to medicine. Numerous studies around the globe are being conducted on the prevention and treatment of this infection. A significant amount of them study the role of vitamin D in the pathogenesis of the disease. Cholecalciferol (Vitamin D) is a fat-soluble vitamin that is involved in maintaining the serum calcium-phosphorus gradient. Vitamin D supplementation significantly reduces the risk of osteoporosis, and also affects the regulation of immune responses by modulating innate and adaptive immune responses. It has been shown to inhibit the proliferation of T cells, namely the subsequent transformation of Th1 cells to Th2 cells. This effect on cell proliferation and differentiation contributes to a significant decrease in the level of proinflammatory cytokines, thereby reducing the severity of immune-mediated damage. It was these mechanisms that formed the basis of the theory about the ability of vitamin D to prevent the severe course of coronavirus infection and even prevent it. At the moment, the effect of vitamin D on reducing COVID-19 morbidity is not fully confirmed.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18 to 75 years
* who did not take Vitamin D supplementation
* COVID-19 clinical features
* signed informed consent to participate in the research.

Exclusion Criteria:

* pregnancy or nursing
* primary hyperparathyroidism or hypercalcemia other etiologies (including 24-hydroxylase mutation)
* a history of granulomatous diseases
* severe gastrointestinal diseases (clinically apparent malabsorption syndrome)
* liver disease
* kidney disease
* individual intolerance drug
* vitamin D supplementation in a dose of more than 800 IU per
* drugs known to affect vitamin D metabolism (e.g., anticonvulsants, glucocorticoids, diuretics)
* alcohol and drug addiction.
* history of cancer (less than 5 years)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Combined: severity, ICU hospitalization, outcome of the disease on 14-21 days | baseline and on 14-21 days
  * Severity of new coronavirus infection- moderate, severe, extremely severe
  * Hospitalization in intensive care unit
  * Outcome of the disease - recovery or fatal outcome

SECONDARY OUTCOMES:
Serum 25(OH)D level | baseline and on 9-10 days
Serum APPs (acute phase proteins) levels, cytokine/chemokine concentrations | baseline and on 14-21 days
  Change in the serum concentration of CRP (C-reactive protein), ferritin, LDH (lactate dehydrogenase), IL-6
Duration of hospitalization | baseline and on 14-21 days
  number of days spent in hospital
Interleukin-6 inhibitors application | baseline and on 14-21 days
  The need to use Interleukin-6 Inhibitors - olokizumab, tocilixamab, levilimab

CONTACTS AND LOCATIONS:
Locations (1):
- Almazov National Medical Research Centre, of the Ministry of Health of the Russian Federation, Saint Petersburg, Russia